CLINICAL TRIAL: NCT06774872
Title: MODULO Trial: Doravirine/Lamivudine (DOR/3TC) as a Maintenance ART in Comparison With Dolutegravir/Lamivudine (DTG/3TC) in PLWH Successfully Treated With Three-drug Regimens at Inclusion
Brief Title: Doravirine/Lamivudine (DOR/3TC) as a Maintenance ART in Comparison With Dolutegravir/Lamivudine (DTG/3TC) in PLWH Successfully
Acronym: MODULO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Collaborators: ANRS, Emerging Infectious Diseases (Other Government); Organization providing support methodology coordination (Institut Pierre Louis d'Epidémiologie et de Santé Publique) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREPATS 19
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — doravirine; Lamivudine; dolutegravir

STUDY DESIGN:
Intervention Model Description: The MODULO trial is a prospective, multicentre, open-label trial, designed to asse the non-inferiority of DOR/3TC, in comparison with DTG/3TC, for maintaining the virological success in PLWH with suppressed viremia under three-drug regimens at inclusion. A follow-up over 96 week is expected.
  The 1:1 randomisation will be centralised and realised by the Methodology and Management Centre. The randomisation will be stratified according to the class of the third antiretroviral agent at time of screening (PI, NNRTI or INSTI), leading to three lists of randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DORAVIRINE/LAMIVUDINE combination (Experimental): Patients randomized to "arm 1" will receive the DORAVIRINE/LAMIVUDINE combination: doravirin (PIFELTRO®) 100 mg 1 tablet per day + lamivudine (generic) 300 mg 1 tablet per day
  The dosage is in accordance with the summary of product characteristics of each product.
  Interventions: Drug: Doravirine 100Mg Tab and Lamivudine 300 Mg Tab
- Fixed DOLUTEGRAVIR/LAMIVUDINE combination (Active Comparator): Patients randomized to arm 2 will receive the fixed combination DOLUTEGRAVIR/LAMIVUDINE: dolutegravir 50 mg/lamivudine 300 mg (DOVATO®) 1 tablet per day.
  The dosage is in accordance with the summary of product characteristics of each product.
  Interventions: Drug: Dolutegravir 50mg Tab and Lamivudine 300 Mg Tab

INTERVENTIONS:
Drug: Doravirine 100Mg Tab and Lamivudine 300 Mg Tab — Participants randomised in the "arm 1" will receive the DORAVIRINE/LAMIVUDINE combination: doravirine (PIFELTRO®) 100 mg 1 pill a day + lamivudine 300 mg 1 pill a day
  Arms: DORAVIRINE/LAMIVUDINE combination
Drug: Dolutegravir 50mg Tab and Lamivudine 300 Mg Tab — Participants randomised in the "arm 2" will receive the DTG/3TC combination: dolutegravir 50 mg/lamivudine 300 mg (DOVATO®) 1 pill a day
  Arms: Fixed DOLUTEGRAVIR/LAMIVUDINE combination

SUMMARY:
The main objective of the MODULO trial is to compare (non-inferiority) the capacity of DOR/3TC and DTG/3TC two-drug regimens of maintain virological success at W48 in people living with HIV virus ( PLWH) with suppressed HIV plasma viral load (pVL) under three-drug regimen at inclusion.

The virological success is defined as no virological failure (2 consecutive pVL ≥50 copies/mL or one pVL ≥50 copies/mL followed with discontinuation of treatment or follow-up).

DETAILED DESCRIPTION:
There is growing interest in antiretroviral therapy for people living with HIV (PLWH) to optimize and reduce the use of antiretroviral treatment (ART). The evaluation of the dual therapies dolutegravir/rilpivirine (DTG/RPV) and dolutegravir/lamivudine (DTG/3TC) in large comparative trials has resulted in their inclusion in international recommendations. EACS and IAS-USA recommend DTG/3TC in patients naïve to treatment. Switch recommendations include more diversified options (DTG/3TC, DTG/PVR, darunavir boosted/lamivudine [DRV/r/3TC]). Recently, injectable intramuscular bicugravir/lamivudine (CAB/RPV) is also available and recommended. Apart from the DRV/r/3TC combination, which has the limitation of being combined with ritonavir, with a lower tolerance and many drug interactions, all these bitherapies rely on integrase inhibitors (INIs).

A significant number of patients cannot benefit from these strategies and their long-term toxicity reduction benefits (due to history of intolerance to certain ARVs, especially INIs, and/or acquired and archived resistance to former non-nucleoside reverse transcriptase inhibitors [INNTIs], including rilpivirine, or INIs), or due to incidental comorbidities, associated with comedyations at risk of drug interactions, accentuated by the aging population of PLHIV.

For this reason, the investigators think it is important to evaluate a new antiretroviral dual therapy that is free of both the use of INIs and the use of boosted IPs.

Also, the combination of an INNTI with lamivudine could fulfill this role. To date, only one pilot study involving 20 patients has evaluated a combination of nevirapine and 3TC. At the 144th week, no virological failure was observed.

Long-term toxicity of ARVs has been well demonstrated for IPs and nucleoside reverse transcriptase inhibitors (INTIs), classes that are widely used in currently treated PHAs. In the French hospital cohort (ANRS-CO4 FHDH), prolonged exposure to IPs was independently associated with an increased risk of myocardial infarction. Exposure to IPs has been associated in other studies with increased lipid parameters (triglycerides, LDL-cholesterol). For INTI, mitochondrial toxicity is likely to be common across the class, although the most important drugs are no longer used. Outside this mitochondrial toxicity, the toxicity of tenofovir disoproxil fumarate (TDF) is the most clearly established. In different cohorts, TDF exposure was associated with bone demineralization (osteogenesis, osteoporosis), partially reversible after treatment discontinuation with a discussed increase in risk of fracture TDF exposure is also associated with an over-risk of impaired renal function. Tenofovir alafenamide (TAF) has been implicated in excess weight gain in several studies and cohorts, independent of associated ARVs. Finally, abacavir has also been associated with increased cardiovascular risk.

Antiretroviral therapy has demonstrated clear short- and medium-term benefits in terms of tolerance, both metabolic, renal and bone. For example, it has been shown that the transition to DTG/RPV or DTG/3TC decreases bone resorption markers and improves renal parameters when TDF is stopped. Or improvement of lipid parameters during the transition to etravirin/raltegravir (ETR/RAL), after the IP has been stopped, or when switching to DTG/3TC, after the TAF +/- of the associated IPs. The long-term and "real life" data are also very reassuring about the durability of bitherapies, and therefore on their good tolerance profile and virological robustness. In the OPERA cohort, treatment discontinuations were less frequent in dual therapy than in triple therapy.

Beyond obtaining and maintaining undetectable plasma viral load, ARV therapy reduces even very slowly the viral reservoir (integrated HIV-DNA), limits systemic inflammation and chronic immune activation and therefore limits associated morbidity, controls viral replication in the anatomical compartments, preventing HIV-related neurological diseases and transmission of the virus from an infected individual to an uninfected individual. The question of the performance of bitherapies in all these areas of observation is regularly raised, and all current scientific data are very reassuring. It was shown that during follow-up, after switching to dual therapy, HIV-DNA levels remained stable compared with continuing triple therapy, as did the proportion of residual CVC.Several sub-groupsStudies have shown that viral replication remains controlled in the neurologic compartment or the seminal compartment under bitherapy. For inflammation, conclusions are more difficult to draw clearly because of the large inter- and intra-individual variability of the markers measured, but no deleterious consequences have been identified so far.

Bitherapies are therefore an option of choice, especially in the context of aging PLWH, which have comorbidities and for whom prevention of toxicities should be a priority. However, due to past intolerances and resistance, already mentioned in the draft, bitherapies based on INIs and INNTIs are not always the best option. Excessive weight gain reported under INI in different clinical trials and cohorts is an argument against universal use of dolutegravir, and this point of discussion is increasingly prominent in consultation. Very recent data suggest that INIs may also be associated with more frequent high blood pressure and diabetes.

Taking advantage of the properties of doravirin, a new generation NNRTI, well tolerated, with a relatively high genetic barrier and a drug interaction profile very close to INIs, the investigators propose to include it in a dual therapy in combination with lamivudine, and to study its ability to maintain virological control.

For all the reasons investigator have just detailed, it seems therefore pertinent to develop a dual therapy without INI, without boosted IP and without rilpivirine in order to be able to adjust the therapeutic proposals to the patients. The combination DOR/3TC seems to us quite relevant in this context.

This trial is to validate the efficacy of the DOR/3TC combination and the study population is not restricted to what could be considered as the "target population" for DOR/3TC dual therapy (patients with intolerances or resistance to ARVs commonly used in current bitherapies).

The main hypothesis, which meets the main objective of the study, is that DOR/3TC dual therapy is able to maintain control of viral replication in PLHIV receiving suppressive triple therapy, and this virological efficacy is not lower than that of the DTG/3TC, S48 and S96 dual therapy.

For the choice of the comparator arm, the investigators opted for DTG/3TC dual therapy. This dual therapy is by far the most widely used today and its virological efficacy has been widely demonstrated. This seems more relevant than proposing the maintenance of a "standard" tritherapy: in this way, all patients included in the study, under tritherapy at inclusion, will benefit from an optimization strategy of ARV treatment, and we will be able to compare the DOR/3TC dual therapy with a reference dual therapy, in terms of virological efficacy and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years;
* Living with HIV-1;
* With pVL <50 copies/mL for at least 24 months;
* Under stable three-drug regimen including 2 NRTIs + 1 NNRTI or 1 INSTI or 1 boosted PI for at least 12 months;
* Affiliated to the French Social Insurance;
* Who have given their written consent to participate in the study

Exclusion Criteria:

* HIV-2 co-infection;
* Co-infection with hepatitis B virus (positive HBsAg and/or positive anti-HBc antibody with negative anti-HBs antibody);
* Documented resistance mutation or association of resistance mutations, associated with partial or full resistance to doravirine, dolutegravir or lamivudine;
* At least one resistance genotype is mandatory to include the patient:

  * If there was no virological failure under NRTI, NNRTI and INSTI in the past:

    * Pretherapeutic HIV-RNA genotype,
    * OR, in case of no available HIV-RNA genotype, genotype on proviral HIV-DNA to performed before inclusion,
  * In case of virological failure under NRTI, NNRTI and INSTI in the past:

    * HIV-RNA genotype at time of virological failure,
    * OR, in case of no available HIV-RNA genotype at time of failure, genotype on proviral HIV-DNA to performed before inclusion to be sure that the virus is fully sensitive to the study treatments,
  * Past virological failure is defined as: 2 consecutive pVL ≥50 copies/mL or one pVL ≥200 copies/mL,
  * Resistance genotypes will be interpretated with the last available ANRS algorithm.
* Glomerular filtration rate <50 mL/min (CKD-EPI formula);
* Comedications leading to drug-drug interaction with one of the 3 study drugs (cf. detailed protocol);
* Pregnant or breastfeeding women, and women with age to be pregnant but refusing effective contraception, whether or not a desire for pregnancy is expressed;
* Any clinal condition limiting the participation in a clinical trial: Immunocompromised conditions including active cancer or hematological malignancy, organ transplant or with transplant rejection within the last 6 months, immunosuppressive therapy, or other condition that in the opinion of the investigator could cause impaired host immunity
* Protected adults (persons under legal guardianship or under "sauvegarde de justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Measure the virological efficacy at week 48 to assess the effectiveness of the dual therapy to maintain the virological success to week 48 | Week 48
  Measure ol plasma viral load assessed by RNA quantification using COBA 6800 system (Roch)

CONTACTS AND LOCATIONS:
Overall Officials: Romain PALICH, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided